CLINICAL TRIAL: NCT05898659
Title: Comparison of a Bimodal Fitting With Synchronization and a Conventional Bimodal Fitting in Newly Implanted Cochlear Patient. Prospective Monocentric Randomized Double-blind Crossover Study.
Brief Title: Comparison in New Cochlear Implanted Subjects of a Tonotopy-based Bimodal Fitting With or Without Synchronization
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: MED_EL_REG_BIMOD_Nice_study
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Sensorineural Hearing Loss, Bilateral
Keywords: cochlear implant; bimodal fitting; tonotopy-based fitting
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Cochlear Implants

STUDY DESIGN:
Intervention Model Description: Two arms A and B:
  Arm A: Bimodal patient's fitting with tonotopy-based fitting without synchronization (ABFnoS) --> 6 weeks use --> tests and bimodal patient's fitting with tonotopy-based fitting with synchronization (ABFS) --> 6 weeks use --> tests; Arm B: Bimodal patient's fitting with ABFS --> 6 weeks use --> tests and bimodal patient's fitting with ABFnoS --> 6 weeks use --> tests
Who Masked: Participant, Investigator
Masking Description: Double blind study: The patient and the investigator don't know the fitting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABFnoS then ABFS (Active Comparator): Cochlear Implant with ABFnoS first during 6 weeks then with ABFS during 6 weeks
  Interventions: Device: ABFnoS then ABFS (Cochlear implant)
- ABFS then ABFnoS (Active Comparator): Cochlear Implant with ABFS first during 6 weeks then with ABFnoS during 6 weeks
  Interventions: Device: ABFS then ABFnoS (Cochlear implant)

INTERVENTIONS:
Device: ABFnoS then ABFS (Cochlear implant) — Cochlear implant with tonotopy-based fitting without synchronization with the contralateral hearing-aid then with synchronization with the contralateral hearing-aid
  Arms: ABFnoS then ABFS
Device: ABFS then ABFnoS (Cochlear implant) — Cochlear implant with tonotopy-based fitting with synchronization with the contralateral hearing-aid then without synchronization with the contralateral hearing-aid
  Arms: ABFS then ABFnoS

SUMMARY:
Main objective:

For a bimodal fitting (hearing aid (HA) + cochlear implant (CI)): Comparison of a tonotopy based fitting strategy with synchronization between HA and CI (ABFS) to a tonotopy based fitting strategy without synchronization (ABFnoS) for the accuracy of sound localization.

Secondary objectives:

Comparison of ABFS to ABFnoS for the bias of sound localization. Comparison of ABFS to ABFnoS for speech perception in noise. Comparison of ABFS to ABFnoS for the auditory skills experienced by the subject.

DETAILED DESCRIPTION:
Introduction: Cochlear implantation allows the rehabilitation of profound bilateral deafness, restoring speech perception and verbal communication when the traditional hearing aid no longer provides satisfactory hearing gain.

A cochlear implant includes an electrode array and its functioning is based on the principle of cochlear tonotopy: Each electrode encodes a frequency spectrum according to its position in the cochlea (high frequencies are assigned to the basal electrodes and low frequencies to the apical electrodes). The cochlear implant thus breaks down the frequency spectrum into a number of frequency bands via bandpass filters corresponding to the number of electrodes in the implant. During the fitting these bands can be modified by the audiologist.

MED-EL has developed a fitting strategy (ABF) that allows, from a post-operative scanner, to calculate the theoretical characteristic frequency of neurons stimulated by each electrode contact and to transmit this information to the fitting software of the CI.

Bimodal hearing refers to the use of a CI in one ear with a HA on the contralateral side.

This association allows for adults and children a better perception of speech in quiet and in noise, a better perception of music, hearing comfort, better sound quality, better localization of sound and, consequently, a better quality of life compared to unilateral CI alone. However, there is great variability in the integration process; while some bimodal users show substantial benefits, others receive little or no benefit.

This variability could be due to different processing times between CI and contralateral HA.

Recently, MED-EL (Austria) has developed a new approach to synchronize the treatment time of the CI with that of the contralateral HA via the fitting software. This new approach takes into account the different treatment times between CI and contralateral HA and allows synchronization between the 2 systems (CI and HA).

This strategy (ABFS) could therefore allow a better integration of information in bimodal hearing and in particular improve the sound localization compare to a strategy without synchronization (ABFnoS).

Main objective:

For a bimodal fitting (hearing aid (HA) + cochlear implant (CI)): Comparison of a tonotopy based fitting strategy with synchronization between HA and CI (ABFS) to a tonotopy based fitting strategy without synchronization (ABFnoS) for the accuracy of sound localization.

Secondary objectives:

Comparison of ABFS to ABFnoS for the bias of sound localization. Comparison of ABFS to ABFnoS for speech perception in noise. Comparison of ABFS to ABFnoS for the auditory skills experienced by the subject.

Plan of the study:

It is a prospective open monocentric randomized crossover study: Measures will be done on the patient at 6 weeks and 12 weeks post-activation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>= 18 years old) speaking French
* Patient who fulfils the criteria for cochlear implantation
* Total hearing loss for less than 5 years

Exclusion Criteria:

* retro-cochlear pathology: auditory neuropathy, vestibular schwannoma
* patient with residual hearing < 70 dB hearing level (HL) at 250 Hz and 500 Hz and < 80 dB HL at 1000 Hz on the contralateral ear

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy of sound localization | at 6 weeks post-activation
  The accuracy of sound localization will be achieved with a sound localization test in the horizontal plane with 7 loudspeakers (HP) spaced 30° apart and arranged in a ½ circle from -90° to +90° at 1m around the patient.
Accuracy of sound localization | at 12 weeks post-activation
  The accuracy of sound localization will be achieved with a sound localization test in the horizontal plane with 7 loudspeakers (HP) spaced 30° apart and arranged in a ½ circle from -90° to +90° at 1m around the patient.

SECONDARY OUTCOMES:
Bias of sound localization | at 6 weeks post-activation
  The bias of sound localization will be achieved with a sound localization test in the horizontal plane with 7 loudspeakers (HP) spaced 30° apart and arranged in a ½ circle from -90° to +90° at 1m around the patient.
Bias of sound localization | at 12 weeks post-activation
  The bias of sound localization will be achieved with a sound localization test in the horizontal plane with 7 loudspeakers (HP) spaced 30° apart and arranged in a ½ circle from -90° to +90° at 1m around the patient.
Speech recognition in noise | at 6 weeks post-activation
  The speech recognition in noise is evaluated with the French-language VRB (vocale rapide dans le bruit) test [Leclerc et al., Eur Ann Otorhinolaryngol Head Neck Dis
  . 2018 Oct;135(5):315-319.]. It is a sentence test with target words. The speech level is at 65 dB sound pressure level (SPL) and the signal-to-noise ratio varies from 18 dB to -3 dB by 3 dB step.
Speech recognition in noise | at 12 weeks post-activation
  The speech recognition in noise is evaluated with the French-language VRB (vocale rapide dans le bruit) test [Leclerc et al., Eur Ann Otorhinolaryngol Head Neck Dis
  . 2018 Oct;135(5):315-319.]. It is a sentence test with target words. The speech level is at 65 dB SPL and the signal-to-noise ratio varies from 18 dB to -3 dB by 3 dB step.
Auditory skills experienced by the patient | at 6 weeks post-activation
  Auditory skills experienced by the patient are evaluated with the French version of the speech spatial qualities scale (SSQ) with of 49 questions describing various real-world auditory situations..
Auditory skills experienced by the patient | at 12 weeks post-activation
  Auditory skills experienced by the patient are evaluated with the French version of the speech spatial qualities scale (SSQ) with of 49 questions describing various real-world auditory situations..

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Guevara, Pr, Principal Investigator — Nice University Hospital
Locations (1):
- CHU Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No